CLINICAL TRIAL: NCT01934517
Title: Validity, Reliability and Reproducibility of Digital Models Obtained With iTero® (AlignTech) and Lava Digital® (3M) in Comparison With Plaster Models.
Brief Title: Validity of Digital Models Obtained With iTero® and Lava Digital® in Comparison With Plaster Models.
Status: Completed | Type: Observational
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Normand Bach, professor, Université de Montréal
Other Study IDs: VCP2013udem
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Dentition/Teeth Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the validity, reliability and reproducibility of digital models obtained from iTero® and Lava Digital® in comparison with traditional plaster models.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the validity, reliability and reproducibility of the dental measurements obtained on the digital models with iTero® in comparison with those obtained on the plaster models (gold standard) and on the digital models with Lava Digital®.

The secondary objective is to compare two different impression materials (i.e. alginate and polyvinylsiloxane (PVS)) and determine whether the impression material used affects the accuracy of the measurements.

Statistical analysis:

* Intraclass correlation coefficient (ICC) will be used to evaluate the intra- and inter-operator reliability of the measurements for each method, i.e. the plaster models and the digital models.
* A paired t-test will be used to determine the validity of the digital measurements with iTero®, and to compare the impression materials (alginate and PVS).
* A Bland-Altman plot will also be used to compare the two digital methods (Lava Digital® et iTero®) with the plaster models.
* Dahlberg coefficient will be used to evaluate the technical error associated with the measurements that will be made.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 30 years old (male or female)
* complete permanent dentition from first molar to the other first molar
* no interproximal modifications (e.g. decay, large restorations, abnormal tooth morphology) which could affect the mesio-distal width of the teeth

Exclusion Criteria:

* Dentition with severe crowding (that could therefore affect the mesio-distal width of the teeth)

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients requiring an orthodontic treatment from the Orthodontics clinic of the University of Montreal
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent-Claude Peloquin, resident, Principal Investigator — University of Montreal, department of Orthodontics; Normand Bach, D.M.D., M.Sc., F.R.C.D.(c), Study Director — Université de Montréal
Locations (1):
- University of Montreal, Faculty of Orthodontics, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- iTero, Lava Digital and Plaster Models: All Study Participants: Single-group study:
  1. ITero models obtained from intraoral scans with iTero scanner
  2. Plaster models obtained from alginate and PVS intraoral impressionsScan of plaster
  3. Lava Digital models obtained from extraoral scans of plaster models
Period: Overall Study
Arm/Group | iTero, Lava Digital and Plaster Models: All Study Participants
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- iTero, Lava Digital and Plaster Models: All study participants: iTero, LavaDigital and plaster models (single-group study)
Arm/Group | iTero, Lava Digital and Plaster Models
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: Overjet
Description: Overjet: measured as the greatest horizontal distance from the labial surface of the lower central incisor to the most inferior point at the mesiodistal center of the upper central incisor
Time Frame: one year
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- iTero Models: ITero models obtained from intraoral scans with iTero scanner
- Plaster Models: Plaster models obtained from alginate and PVS intraoral impressionsScan of plaster
- Lava Digital Models: Lava Digital models obtained from extraoral scans of plaster models
Arm/Group | iTero Models | Plaster Models | Lava Digital Models
Number analyzed (Participants) | 25 | 25 | 25
mm | 0.25 [-0.65 to 1.16] | 0.27 [-0.78 to 1.25] | 0.28 [-0.58 to 1.20]

ADVERSE EVENTS:
Arm/Group | iTero Models | Plaster Models | Lava Digital Models
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No